CLINICAL TRIAL: NCT00204230
Title: Randomized Controlled Study: Effect of Mycophenolatmofetil in Patients With Histologically Proven Chronic Allograft Nephropathy
Brief Title: MMF and Calcineurin Inhibitor Withdrawal in CAN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Immunosuppressive Agents; Kidney Failure, Chronic; Kidney Transplantation
Keywords: Kidney Failure, Chronic; Kidney Transplantation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Mycophenolic Acid; Pharmaceutical Preparations

INTERVENTIONS:
Drug: mycophenolate mofetil (drug)

SUMMARY:
Prospective, randomised study: Effect of mycophenolatmofetil (MMF) and CNI withdrawal in patients with histologically proven chronic allograft nephropathy Indication: change in immunosuppressive treatment of chronic allograft nephropathy (CAN)after renal transplantation Hypothesis: Antimetabolite MMF is able to stop progression of CAN and improve blood pressure/ metabolic parameters and structural vessel wall changes

Primary Target:effects of CNI withdrawal and MMF on renal function: stabilisation and/or improvement Secondary Targets: Incidence of adverse events Evaluation of the calcineurin inhibitor free MMF treatment effects on blood pressure, lipids, glucose metabolism and on structural and functional vesselwallchanges Method:open prospective, randomized two-tailed, monocentric study

DETAILED DESCRIPTION:
Prospective, randomised study: Effect of mycophenolatmofetil in patients with histologically proven chronic allograft nephropathy

SYNOPSIS

Indication: change in treatment to improve the course of chronic allograft nephropathy

Method: open prospective, randomized two-tailed, non blinded monocentric study

Follow up period: 35 Weeks

Number of patients: 2 x 86 patients

Inclusion criteria: • Written informed consent

* Reduction of graft function: Increase of serum creatinine >/= 0,1mg/dl/month in the previous 6 months before start of the study and/or new occurrence or increasing proteinuria in the last 6 months before start of the study
* Serum creatinine < 4 mg/dl
* Biopsy within the last 3 months
* histologically proved chronic allograft nephropathy (graft glomerulopathy, chronic rejection ,interstitial fibrosis, tubular atrophy, vascular arteriosclerosis,hyalinosis)
* >1 year after renal allografting
* At least 5 mg/day of prednisolone or equivalent dose

Exclusion criteria: • Malignomas

* Gravidity or Lactation
* Participation in other studies
* Severe infections
* Florid gastrointestinal Ulcer
* Age between 18 and 70 years
* Leukopenia with less that 3000/l leucocytes, Anaemia Hb  9 g/dl
* Therapy with mycophenolatmofetil in the past 6 months
* Acute rejections in the apst 6 months

Study protocol:

Phase I: Week 1.-3. Conversion to Triple-Drug-Therapy, consisting of Mycophenolatmofetil, corticosteroids (e.g. prednisolone) and ciclosporine A or Tacrolimus

1. Addition of Mycophenolatmofetil (MMF) to the previous immosuppressive treatment, consisting of ciclosporine A (CsA) or Tacrolimus (FK506) in combination with corticosteroids, e.g. prednisolone (P). In the case that azathioprine (AZA) had been given, AZA is replaced by MMF. The therapy with MMF starts 3 days after the elimination of azathioprine.

The addition of MMF follows the following scheme if nothing else is indicated:

1. week: 1g/day, 2.week: 1,5g/day, 3.week: 2g/day
2. Ciclosporine A bzw. tacrolimus: Target whole trough blood levels:

   CsA: 80-120 ng/ml (HPLC) FK506: 4-7 ng/ml (IMX Tacrolimus, Abbott)
3. Corticosteroids, e.g. prednisolone: The previous dosage is continued, but at least 5 mg prednisolone/day (or equivalent) must be given

Phase II: week 4.-9.

Randomisation at the beginning of week 4:

All patients receiving at least 3 x 500 mg MMF per day were randomised as follows Group A: Continuation of the triple therapy Group B: Elimination of CsA bzw. FK506 The ciclosporine A- or tacrolimus-dosage is reduced ba 33% each 2 weeks so that after 6-8 weeks a total elimination of the drugs is reached.

Phase III: week 10.-35.

Continuous therapy with...:

Group A: Triple therapy MMF / CsA bzw. FK506 / Corticosteroids e.g. Prednisolone Group B: Dual therapy MMF / Corticosteroids e.g. Prednisolone

Primary Endpoint:

Comparison of the development of 1/creatinine in both branches 32 weeks after randomization

Secondary Endpoints:

* Occurrence of...

  * acute rejections
  * infections
  * malignomas
  * gastrointestinal disorders
* Blood pressure evolution and number of antihypertensive drugs
* Changes concerning the lipid state
* Changes concerning the glucose metabolism
* Changes in metabolism of uric acid
* Comparison of the development of 1/creatinine within each branch 6 months before and 6 months after therapy conversion
* Comparison of drop out rate in branches A und B
* Pharmacokinetics of mycophenolic acid (MPA) based on a new method of abbreviated area under the curve (AUC) determination
* vessel wall changes of the carotid arteries measured by high resolultion ultrasound methods and hemodynamic parameters measured by task force equipment before and 9 month after cni withdrawal and MMF addition

Criteria for study discontinuation:

* Sepsis
* Occurrence of acute rejections
* Graft loss
* Other severe adverse events
* patients decision

ELIGIBILITY:
Inclusion Criteria:

Written informed consent Reduction of graft function: Increase of serum creatinine >= 0,1mg/dl/month in the previous 6 months before start of the study and/or new occurrence or increasing proteinuria in the last 6 months before start of the study Serum creatinine < 4 mg/dl Biopsy within the last 3 months histologically proved chronic allograft nephropathy >=1 year after renal allografting >=5 mg/day Prednisolone or equivalent dose

Exclusion Criteria:

Malignomas Gravidity or Lactation Participation in other studies Severe infections gastrointestinal Ulcer Age <18 and >70 years Leukopenia with less that 3000/dl leucocytes, Anaemia Hb > 9 g/dl Therapy with mycophenolatmofetil in the past 6 months Acute rejections in the past 6 months

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Start 1999-10; Study Completion 2002-09

PRIMARY OUTCOMES:
course of renal function over 35 weeks

SECONDARY OUTCOMES:
after 35 weeks of follow up:
incidence of
-acute rejections
-infections
-malignomas
-gastrointestinal disorders
development of blood pressure over 35 weeks
number of antihypertensive drugs
lipid state at entry and after 35 weeks
blood glucose ,HBA1c at entry and after 35 weeks
uric acid at entry and after 35 weeks
Comparison of the development of 1/creatinine within each group at entry and 35 weeks after therapy conversion
area under the curve (AUC) determination of mycophenolic acid (MPA)
vessel wall changes of the carotid arteries IMD , compliance, distensibility and hemodynamic parameters CO, CI, at entry and after after cni withdrawal and MMF addition

CONTACTS AND LOCATIONS:
Overall Officials: Barbara M Suwelack, PhD, Principal Investigator — University Hospital

REFERENCES:
- [Result] Suwelack B, Gerhardt U, Hohage H. Withdrawal of cyclosporine or tacrolimus after addition of mycophenolate mofetil in patients with chronic allograft nephropathy. Am J Transplant. 2004 Apr;4(4):655-62. doi: 10.1111/j.1600-6143.2004.00404.x. PMID 15023160